CLINICAL TRIAL: NCT03325946
Title: The FBRI VTC Neuromotor Research Clinic
Status: Recruiting | Type: Observational
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Stephanie DeLuca, Associate Professor, Virginia Polytechnic Institute and State University
Other Study IDs: 13-196
Record Dates: First submitted 2017-10-09; First posted 2017-10-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Neuromotor Impairments; Cerebral Palsy; Microcephaly; Autism; Trauma, Brain; Acquired Brain Injury; Pediatric Stroke
MeSH Terms: conditions — Cerebral Palsy; Microcephaly; Autistic Disorder; Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children and Adults with Cerebral Palsy
  Interventions: Behavioral: ACQUIRE Therapy
- Children and Adults with Microcephaly
  Interventions: Behavioral: ACQUIRE Therapy
- Children and Adults with other Neuromotor Impairments
  Interventions: Behavioral: ACQUIRE Therapy
- Children who have had a stroke
  Interventions: Behavioral: ACQUIRE Therapy

INTERVENTIONS:
Behavioral: ACQUIRE Therapy — Intensive therapy services combined with operant conditioning during treatment delivered by trained OT or PTs

SUMMARY:
The FBRI VTC Neuromotor Research Clinic was established and opened in May of 2013 to provide intensive therapeutic services to individuals with motor impairment secondary to neuromotor disorders. It is direct by Dr. Stephanie DeLuca and based on the principles surrounding ACQUIREc Therapy.

ACQUIREc Therapy is an evidenced-based approach to pediatric constraint-induced movement therapy, which refers to a multi-component form of therapy that is focused on helping children who have asymmetric motor abilities between the two sides of the body. Historically, ACQUIREc Therapy has the unimpaired or less impaired upper extremity constrained (by a cast or a splint) while also receiving active therapy from a specially trained therapist who shapes new skills and functional activities with the child's more impaired upper extremity but who is also a licensed Occupational or Physical Therapist (OT/PT). Therapy dosages are high much higher than tradition OT or PT - often lasting many hours per day, up to 6 hours a day, 5 days a week, for 2-4 weeks.

Investigators have developed further treatments based on the same principles of intensive services combined with behavior shaping for other areas of the body that are also affected by weakness (e.g., the leg and trunk) also, but which usually do not involve constraint. These have been more generally labeled ACQUIRE Therapy.

All forms involve intensive, play-based therapy for children with asymmetric motor impairments of the arms and hands. The primary focus of treatment is to facilitate the acquisition of new motor skills in the child's weaker body parts through high levels of intensive therapy using scientifically-based behavioral guidelines. Therapy is also delivered in naturalistic environments.

ACQUIREc Therapy as a treatment method has been tested in two randomized controlled trials, and a specific manual for its implementation has been developed. Dr. (s) Ramey and DeLuca previously founded a similar clinic, The Pediatric Neuromotor Research Clinic, at the University of Alabama at Birmingham where Dr. DeLuca directed the research clinic for 13 years and oversaw the implementation of the ACQUIREc Therapy treatment protocol in more than 400 cases.

This research will involve analyzing and interpreting the clinical data of children going through clinical procedures at the FBRI VTC Neuromotor Research Clinic. All participation is voluntary and no children will denied services if families choose not to participate.

ELIGIBILITY:
Inclusion Criteria:

* Neuromotor Impairment

Exclusion Criteria:

* fragile health

Ages: 3 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Individuals with neuromotor impairment who want to try and gain motor skills and function
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Emerging Behaviors Scale | up to 12 months
  This is a measure of the number of skills a child uses from a set of 31 typical used on a daily basis

SECONDARY OUTCOMES:
Assisting Hand Assessment | Within 1 week prior to treatment and Within 1 week after treatment
  This is a measure of bimanual arm and hand use
Pediatric Motor Activity Log | Within 1 week prior to treatment and Within 1 week after treatment
  This is a parental report about a child's ability to use an impaired arm and hand on a daily basis
Peabody Developmental Motor Scales 2 | Within 1 week prior to treatment and Within 1 week after treatment
  This is a measure of a child's motor abilities in comparison to typical development
The Bayley Motor Scales of Infant Development -III | Within 1 week prior to treatment and Within 1 week after treatment
  This is a measure of a infants's motor abilities in comparison to typical development

OTHER OUTCOMES:
Video Assessments | Within 1 week prior to treatment, during treatment, and Within 1 week after treatment
  Videos of play and therapy sessions

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie DeLuca, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Fralin Biomedical Research Institute - VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Data is released only with participant (parental/ guardian) permission

REFERENCES:
- [Derived] Wallace DA, Rebekah Trucks M, DeLuca SC. Clinical use of ACQUIRE Therapy for Children Diagnosed With CASK-Gene Related Disabilities. Adv Rehabil Sci Pract. 2024 Nov 27;13:27536351241302852. doi: 10.1177/27536351241302852. eCollection 2024 Jan-Dec. PMID 39610761
- [Derived] DeLuca SC, Wallace DA, Trucks MR, Mukherjee K. A clinical series using intensive neurorehabilitation to promote functional motor and cognitive skills in three girls with CASK mutation. BMC Res Notes. 2017 Dec 19;10(1):743. doi: 10.1186/s13104-017-3065-z. PMID 29258560